CLINICAL TRIAL: NCT00463671
Title: The Relation Between Hyperbaric Oxygen, Oxidative Stress, NO Bioavailability and Tissue Oxygenation in Diabetic Patients Suffering From Foot Ulcers
Brief Title: Hyperbaric Oxygen, Oxidative Stress, NO Bioavailability and Tissue Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HBO2/03
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-05

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: N-acetylcysteine

SUMMARY:
Hyperbaric oxygen therapy (HBOT) increases tissue oxygenation and serves as an adjunct therapy for diabetic wounds. However, some patients have insufficient increase or even paradoxical decrease in tissue O2 due to vasoconstriction. The aim of the present study was to investigate the pathophysiology responsible for the different consequences of HBOT and to evaluate the effect of N-acetylcysteine (NAC) on these changes.

Methods: Prospective, randomized, cross-over trial including fifty diabetic patients with non-healing ulcers. All patients had two HBOT (100%oxygen, 2ATA) with NAC at the first or the second evaluation. At the beginning and at the end of each evaluation, ulcer oxygenation and plasma levels of malondialdehyde (MDA), total anti-oxidant status (TAOS) and nitric oxide (NO) were measured. Patients with ulcer oxygenation above 200mmHg, were subjected to complete HBOT protocol.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients, aged 18 years or older, with non-healing foot ulcers

Exclusion Criteria:

* Patients with macrovascular disease amenable for revascularization with more than 70% obstruction in femoral artery (evaluated by US doppler) were excluded from the study. Similarly, patients with a documented allergy to NAC, liver cirrhosis or those receiving NAC for other indications were excluded. Finally, patients with chest pathology incompatible with pressure changes, patients with inner ear disease, or those suffering from claustrophobia were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-12; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The aim of the present study was to investigate whether changes in oxidative stress and NO bioavailability are responsible for the different effects of HBOT on tissue oxygenation in diabetic patients suffering from foot ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- The Institute of Hyperbaric Medicine and Wound Care Clinic, Ẕerifin, Israel